CLINICAL TRIAL: NCT05531604
Title: Appetitive Conditioning in Anorexia Nervosa: Neural, Physiological, and Behavioral Mechanisms
Brief Title: Appetitive Conditioning in Anorexia Nervosa
Acronym: ACAN
Status: Recruiting | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Southern California (Other); University of Toronto (Other); California Institute of Technology (Other); Klarman Family Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20202201
Record Dates: First submitted 2022-08-30; First posted 2022-09-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa
Keywords: appetitive conditioning; pavlovian conditioning; reward learning; reinforcement learning; associative learning; extinction
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AN-Restricting (AN-R): Meet Diagnostic and Statistical Manual (DSM-5) criteria for anorexia nervosa, restricting subtype
  Interventions: Behavioral: appetitive conditioning
- Weight Restored AN-Restricting (WRAN-R): * History of anorexia nervosa, restricting type - previously meeting full DSM-5 criteria.
  * Eating Disorder Examination Questionnaire (EDE-Q) ≤ 2 (within 1 standard deviation [SD] of community norms and lower than 1 standard deviation from clinical norms for female anorexia nervosa, restricting type populations)
  Interventions: Behavioral: appetitive conditioning
- Healthy controls: Healthy females from any racial or ethnic background, not meeting DSM-5 criteria for any psychiatric disorder.
  Interventions: Behavioral: appetitive conditioning

INTERVENTIONS:
Behavioral: appetitive conditioning — The investigators will examine acquisition and extinction of learned associations to positively-valenced, socially rewarding yet symptom-neutral infant laughter sounds in an appetitive conditioning paradigm. The investigators will also examine spontaneous recovery of this association 24 hours later when re-presented with these cues, and the reinstatement of this association when re-exposed to infant laughter.

SUMMARY:
Anorexia nervosa (AN) is characterized by a reduced drive to pursue rewarding experiences and stimuli. Food consumption - which is almost universally experienced as pleasurable - is not described as rewarding by those with AN. This is thought to be underpinned by abnormalities around reward learning. However, the most fundamental question relating to reward in AN - whether those with AN may learn positive associations - remains unaddressed.

In this study, the investigators will identify the patterns of how those with AN acquire positive associations, how they diminish, and their relationships to physiology (heart rate and pupil responses) and brain activation. In assessing the robustness of this learning, the investigators will investigate the extent to which this association is reactivated after 24 hours, and the extent to which a memory prompt will help reinstate this previously learned positive association.

This project will allow for important advances in our understanding of the neurobiology of AN. The investigators will first identify if, and how, those with AN come to learn positive associations to cues, and secondly, the extent to which learned positive associations remain over time. Moreover, the investigators will use machine learning to ascertain whether reward learning can be predicted by physiological and neural biomarkers.

DETAILED DESCRIPTION:
Individuals with anorexia nervosa (AN) suffer from anxiety, reduced pleasure from normally rewarding situations (anhedonia), and disturbed body image. However, restriction of calories from their morbid fear of weight gain, resulting in starvation, typically brings them to attention and has been the primary focus of most treatments and many research studies. Yet, treatments have largely been inadequate, with remission rates less than 25%. Anhedonia and disturbances in reward may be important targets of new treatment approaches. Those with AN report little pleasure in food consumption, social domains, and pursuit of novelty and fun. Neuroimaging studies demonstrate disturbances in reward circuits in response to food- and body-related stimuli and monetary rewards, but results are inconsistent. This may be due to confounding effects of anxiety triggered by symptom-related stimuli. Further, a fundamental process of the overall reward response that has not been studied in AN is reward learning - how one's brain learns to associate stimuli with the experience of reward ("appetitive Pavlovian conditioning"). To investigate this, the investigators will enroll 30 underweight individuals with AN, 30 with weight-restored AN, and 30 healthy controls ages 12-22 to perform a reward conditioning paradigm. The investigators will use infant laughter, a social reward with robust effects that is unlikely to be confounded by other co-occurring symptoms. To understand associated neural activity and physiological responses, the investigators will perform conditioning and examine reinstatement 24-hours later, while obtaining functional magnetic resonance imaging, heart rate deceleration, and pupil dilation data, in addition to subjective degrees of positive experience. Data from underweight and weight-restored AN will further allow us to probe starvation state-related effects. Results will advance our understanding of how reward stimuli are learned and the associated aberrant neural or physiological markers. This will yield a comprehensive mechanistic understanding of hedonic functioning in AN to rationally inform future novel treatment development.

ELIGIBILITY:
Inclusion Criteria:

1. AN-Restricting (AN-R) Group

   Inclusion criteria:
   1. Females from any racial or ethnic background
   2. Ages between 12 and 22 years
   3. Meet DSM-5 criteria for AN - restricting subtype
   4. Medically stable designated by their physician in the past month (having any of the following measurements taken by a physician or nurse within the past month preceding the telephone screen: (i) orthostasis: drop in systolic blood pressure > 20 mm Hg or diastolic blood pressure > 10 mm Hg, or an increase in heart rate (HR) > 20 bpm upon standing for 3 minutes after lying down; (ii) resting HR <45; or (iii) resting blood pressure of <80 mm Hg systolic or <50 mm Hg diastolic 99. Prospective participants who do not meet the medical instability criteria and otherwise pass the telephone screen, will be invited to proceed to the consent process. If they have not had these measurements done in the month prior, we will encourage them to visit their doctor or nurse to have these done and then to recontact us with the results ):
   5. BP and pulse measured at the day of the scan by the investigators

      * Heart rate ≥ 45 at rest
      * Resting blood pressure of ≥80 mm Hg systolic and ≥50 mm Hg diastolic
      * Lying and standing (after 3 min.) BP drop of ≤20 systolic and ≤10 diastolic and increase in HR ≤20 bpm
   6. Not taking psychiatric medications or taking serotonin-reuptake inhibitor or serotonin-norepinephrine reuptake inhibitor medications at stable doses
2. History of AN-Restricting Group:

   Inclusion criteria:
   1. Females from any racial or ethnic background
   2. Ages between 12 and 22 years
   3. EDE-Q ≤ 2 (puts them within 1 standard deviation [SD] of community norms and lower than 1 SD from clinical norms for female AN-R)
   4. History of AN - meeting full criteria, diagnosed by a licensed clinician
   5. Not taking psychiatric medications or taking serotonin-reuptake inhibitor or serotonin-norepinephrine reuptake inhibitor medications at stable doses
3. Healthy controls:

Inclusion criteria:

1. Healthy females from any racial or ethnic background
2. Ages 12-22 years

Exclusion Criteria:

* AN-R and History of AN-R groups:

  1. Antipsychotic medications
  2. Change in dose of psychotropic medication over the previous 4 weeks
  3. Current psychotic disorder

Healthy controls:

1. Any current Axis I disorder
2. Eating Disorder Examination Questionnaire score greater than established community norms (>2)
3. Met criteria for AN (in the past or present)

All:

1. Neurological disorder
2. Infants or children of their own
3. Pregnancy
4. Current risk of suicide with a plan and intent
5. Ferromagnetic metal implantations or devices (electronic implants or devices, infusion pumps, aneurysm clips, metal fragments or foreign bodies, metal prostheses, joints, rods or plates)

Ages: 12 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — We will ask participants to report their identified gender.
Study Population: Investigators will enroll 90 female participants between the ages of 12 and 22 (30 with current anorexia nervosa - restricting type, 30 with a history of anorexia nervosa - restricting type, and 30 non-clinical healthy controls).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Positive valence | Day 1
  A 10-point Likert scale will assess self-reported pleasantness and arousal for each conditioned stimulus, and unconditioned stimulus expectancy
Positive valence | Day 2
  A 10-point Likert scale will assess self-reported pleasantness and arousal for each conditioned stimulus, and unconditioned stimulus expectancy
Pupillary dilation | Day 1
  Measured with an eye-tracking camera
Pupillary dilation | Day 2
  Measured with an eye-tracking camera
Heart rate deceleration | Day 1
  Measured with an electrocardiogram
Heart rate deceleration | Day 2
  Measured with an electrocardiogram
Brain activation | Day 1
  Neural activation in reward circuits measured with functional magnetic resonance imaging
Brain activation | Day 2
  Neural activation in reward circuits measured with functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Feusner, M.D., Principal Investigator — Centre for Addiction and Mental Health; Stuart Murray, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray SB, Zbozinek TD, Craske M, Tadayonnejad R, Strober M, Bari AA, O'Doherty JP, Feusner JD. Neural, physiological, and psychological markers of appetitive conditioning in anorexia nervosa: a study protocol. J Eat Disord. 2022 May 10;10(1):68. doi: 10.1186/s40337-022-00546-5. PMID 35538507
- See also: Published manuscript of the study protocol — https://jeatdisord.biomedcentral.com/articles/10.1186/s40337-022-00546-5